CLINICAL TRIAL: NCT05818709
Title: A Multicenter, Evaluator-blinded, Randomized, Delayed Treatment Control Study of the Safety and Effectiveness of HAC 22L for Improving Midface Volume
Brief Title: A Study to Assess Adverse Events and Effectiveness of HAC 22L Injection for Mid-Face Volume in Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M21-846
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Facial Volume Deficit
Keywords: Mid-Face Volume; HAC 22L; VOLUMIZE

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HAC 22L (Experimental): Participants will be randomized to receive HAC 22L on Day 1. Participants will have the opportunity to receive optional touch-up and optional repeat treatment of HAC 22L during the follow-up period.
  Interventions: Device: HAC 22L
- Control Group (Other): Participants can opt to receive HAC 22L after a control period of 6 months. Participants will have the opportunity to receive an optional touch-up treatment and will be followed for an additional 6 months period.
  Interventions: Device: HAC 22L

INTERVENTIONS:
Device: HAC 22L — Subcutaneous and/or Supraperiosteal injection

SUMMARY:
Collagen, elastin, and glycosaminoglycans, (eg, hyaluronic acid) are predominant component of the skin and they are key contributor to its characteristics such as strength, elasticity, and plumpness. Chronic reduction in any one of these components as well as a loss of muscle and fat mass contribute to the facial volume loss that characterizes the aging face. HAC 22L is a dermal filler administered via subcutaneous/supraperiosteal injection for volumizing effect. The purpose of the study is to assess adverse events and effectiveness of HAC 22L in adults with facial volume deficit.

HAC 22L is a novel injectable device being developed to improve mid-face volume. Participants are placed in 1 of 2 groups, called treatment arms. There is a 1 in 3 chance that participants will be assigned to the control group. Around 75 adult participants seeking improvement of mid-face volume will be enrolled in the study at approximately 20 sites worldwide.

Participants in the treatment group will receive HAC 22L injection at Day 1. Participants will have the opportunity to receive optional touch-up and will be followed for up to 24 months. An optional repeat treatment will be offered after the follow-up period. Participants in the control group will followed for 6 months (no treatment period). At completion of the control period, participants may exit or opt to receive the study treatment (inclusive of optional touch-up). Participants will then be followed for 6 months. No repeat treatment is offered to the control group.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by different methods such as medical assessments, questionnaires and instrument's measures.

ELIGIBILITY:
Inclusion Criteria:

* Participant in general good health
* Seeking improvement/correction of mid-face volume
* Participant has overall mid-face severity of Moderate (3), Significant (4), or Severe (5) on the 6-point photonumeric MFVDS as assessed by the EI
* Participant capable of giving signed informed consent

Exclusion Criteria:

* Has experienced trauma to the mid-face within 6 months before enrollment or has residual deficiencies, deformities, or scarring.
* Conditions that could interfere with device effectiveness such as current cutaneous or mucosal inflammatory or infectious processes (eg, herpes), rosacea, abscess, an unhealed wound, active acne, or a cancerous or precancerous lesion in the mid-face
* History of keloid scar formation, hypertrophic scarring, and/or post inflammatory hyperpigmentation
* History of pigmentation disorders or current pigmentation disorder in the face
* A history of facial surgeries in the mid-face
* Received fat injection or permanent implants (eg, polymethylmethacrylate, silicone, polytetrafluoroethylene) anywhere in the face, or is planning to be implanted with any of these products at any time during the study
* Received semipermanent soft-tissue filler treatment (eg, calcium hydroxyapatite, poly-L-lactic acid) in the mid-face within 36 months before enrollment, or is planning to be implanted with any of these products at any time during the study
* Temporary soft tissue filler injections in the mid-face within 24 months before enrollment
* Received botulinum toxin treatment to the midface within 6 months before enrollment, or is planning to undergo any such treatment during the study
* Received mesotherapy or cosmetic facial procedures in the mid-face within 6 months before enrollment, or is planning to undergo any such treatment during the study
* Any over-the-counter or prescription oral or topical, anti-wrinkle products for the mid-face within 30 days before enrollment (participants who have been on a regimen of such products for at least 30 days are eligible for the study if they intend to continue their regimen throughout the study)
* Is on a prescribed regimen of anti-coagulation therapy (eg, warfarin, clopidogrel)
* Tattoos, piercings, hair, or scars that would interfere with visualization of the cheek area for the effectiveness assessments
* Pregnant, nursing, or planning a pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-12-05 (Actual); Study Completion 2025-12-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status Based on the Evaluating Investigator's (EI) live assessment of Mid-Face Volume Deficit Scale (MFVDS) | Month 6
  A "responder" is a participant with at least 1- grade improvement (reduction) of mid face soft tissue deficit using the MFVDS. MFVDS is a validated 6-point scale (0 = None, 5 = Severe).
Number of Participants with Adverse Events | Up to approximately 25 Months
  An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a study intervention which does not necessarily have a causal relationship with the treatment. The investigator assesses the relationship of each event to the use of the study intervention.

SECONDARY OUTCOMES:
Change from baseline on the Rasch transformed score of the FACE-Q Satisfaction with Cheeks module | Month 6
  In the FACE-Q Satisfaction with Cheeks questionnaire, the responses will be summed and converted to a Rasch transformed score that ranges from 0 to 100.
Percentage of Participants Achieving "Responder" Status based on Evaluating Investigator (EIs) assessments of Global Aesthetic Improvement in the treatment area using the Global Aesthetic Improvement Scale (GAIS) | Month 6
  A "responder" is a participant who achieves "Improved" or "Much Improved" on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the cheek area (2=Much Improved, -2=Much Worse).
Percentage of Participants Achieving "Responder" Status based on Participant's assessments of Global Aesthetic Improvement in the treatment area using GAIS | Month 6
  A "responder" is a participant who achieves "Improved" or "Much Improved" on GAIS. GAIS is a 5-point scale used to assess global aesthetic improvement of the cheek area (2=Much Improved, -2=Much Worse).

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (17):
- Germany (11):
  - Hautok and Hautok-cosmetics /ID# 243800, Munich, Bavaria
  - Dermatologie Mahlow /ID# 243805, Blankenfelde-Mahlow, Brandenburg
  - Haut- und Lasercentrum Potsdam /ID# 243822, Potsdam, Brandenburg
  - Rosenpark Research /ID# 243804, Darmstadt, Hesse
  - MediCorium Zentrum fuer Dermatologie und Aesthetik /ID# 243799, Oberursel, Hesse
  - Hautarztpraxis Dr. Niesmann und Dr. Othlinghaus /ID# 243802, Bochum, North Rhine-Westphalia
  - Hautzentrum Koeln /ID# 244607, Cologne, North Rhine-Westphalia
  - Privatpraxis Dr. Hilton & Partner /ID# 243798, Düsseldorf, North Rhine-Westphalia
  - Universitaet Hamburg /ID# 251970, Hamburg
  - Noahklinik GmbH /ID# 244610, Kassel
  - Privatpraxis fuer Dermatologie und Aesthetik /ID# 243803, München
- Spain (6):
  - Instituto Medico Miramar /ID# 251640, Málaga, Malaga
  - Antiaging Group Barcelona (AGB) /ID# 245446, Barcelona
  - Instituto de Medicina y Dermatologia Avanzada (IMDA) /ID# 243339, Madrid
  - Sclinic /Id# 243340, Madrid
  - Grupo Pedro Jaen /ID# 243347, Madrid
  - Instituto de Dermatologia Integral (IDEI) /ID# 245764, Madrid

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-846